CLINICAL TRIAL: NCT02480478
Title: Diagnostic Accuracy of Serum Autotaxin Levels in Cholestasis of Pregnancy
Brief Title: Serum Autotaxin Levels in Cholestasis of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hakan Erenel, MD, OB/GYN, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 518
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: Intrahepatic Cholestasis of Pregnancy
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 5ml whole blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intrahepatic cholestasis of pregnancy: 5 ml whole blood sample is going to collect from intrahepatic cholestasis of pregnancy group for the assessment of serum autotaxin levels
- healthy control group: 5 ml of whole blood is going to taken from healthy control group

SUMMARY:
Intrahepatic cholestasis of pregnancy is the most common liver disease in pregnancy. It is is a pregnancy-specific liver disorder with onset mainly in the third trimester of pregnancy. ICP is characterized by pruritus, elevated serum fasting bile salts and transaminases and an increased risk of adverse fetal outcomes. Serum autotaxin levels were found highly sensitive and specific biomarker to to differentiate ICP from other pregnancy-related liver disorders or pruritic dermatoses. The purpose of the study is to determine the diagnostic accuracy of serum autotaxin activity in cholestasis of pregnancy.

DETAILED DESCRIPTION:
Collected data will enable us to compare serum autotaxin levels in cholestasis of pregnancy and healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed cholestasis of pregnancy patients

Exclusion Criteria:

* acute or chronic liver disease
* acute or chronic gallbladder disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who are admitted to obstetrics and gynecology department due to cholestasis of pregnancy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Serum autotaxin levels in cholestasis of pregnancy | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Erenel, MD,OBGYN, Study Director — Sisli Etfal Training and Research Hospital
Locations (1):
- Sisli Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)